CLINICAL TRIAL: NCT00346021
Title: Sun Protection for Florida's Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Roetzheim, Professor of Family Medicine, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA103965-01 (NIH)
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Skin Cancer
Keywords: Children's behavior towards hat use
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sun Protection Intervention (Experimental): School based sun protection education, provision of free hats.
  Interventions: Behavioral: Increasing hat use
- Control arm (No Intervention): Usual sun protection practices

INTERVENTIONS:
Behavioral: Increasing hat use — Sun protection intervention that address sun protection knowledge, attitudes, social norms, and perceived behavioral controls. Intervention also provides free wide brimmed hats
  Arms: Sun Protection Intervention

SUMMARY:
Purpose of the project is to develop a school-based intervention aimed at increasing hat use when children are outside at home and at school. The intervention is targeted to fourth grade children in Hillsborough County, Florida and is based on Theory of Reasoned Action and Planned Behavior. It is structured to accomplish the following goals: (a) increase sun protection knowledge of children in regards to hat use,(b) foster more positive attitudes in regard to wearing hats,(c) change the subjective norms of wearing hats (d) target persons that children perceive as controlling their behavior of wearing hats(parents,teachers) and increase the use of hats when children are outdoors at school(primary outcome) and when outdoors at times other than school(secondary outcome).

DETAILED DESCRIPTION:
Intervention is aimed at encouraging students to use a wide brim hat when participating in outdoor activities. To accomplish this goal our approach will be multifaceted and will include:

1. individual sessions with school principals to facilitate a school policy that encourages hat use when children are outdoors.
2. sessions with fourth grade teachers that explains the importance of sun protection and hat use, and that addresses potential concerns by teachers.
3. classroom sessions with fourth grade children that improves sun protection knowledge, fosters more positive attitudes about hat use. and that changes the subjective norm of wearing hats when at school.
4. follow-up sessions in which children are provided free hats with a customized design that represents their school.
5. sun protection educational materials that are mailed to the parents of targeted children.

ELIGIBILITY:
Inclusion Criteria:

* One fourth/one fifth grade class.
* 20 students minimum.
* 25% of students are Caucasian.
* Principle/teachers agree to participate.
* Majority of parents agree to participate.
* Majority of 4th grade students provide written assent.
* One outdoor session lasting 20 minutes once per week where children are directly exposed to the sun.
* Outdoor session in an area observable by data monitors.
* School can accommodate intervention components of study.
* School environment stable over the intervention period.
* Randomized control school delay sun protection initiatives until project is completed.

Exclusion Criteria:

-

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2984 (Actual)
Dates: Start 2005-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Increase the use of hats when children are outside at school | june 2008

SECONDARY OUTCOMES:
Increase the hat use when children are outside at times other than school | june 2008

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Roetzheim, MD, MSPH, Principal Investigator — Department of Family Medicine, USF
Locations (1):
- Univeristy of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Roetzheim RG, Love-Jackson KM, Hunter SG, Lee JH, Chen R, Abdulla R, Wells KJ. A cluster randomized trial of sun protection at elementary schools. Results from year 2. Am J Prev Med. 2011 Dec;41(6):615-8. doi: 10.1016/j.amepre.2011.08.005. PMID 22099239
- [Derived] Hunter S, Wells KJ, Jacobsen PB, Lee JH, Boulware D, Love-Jackson K, Abdulla R, Roetzheim RG. Assessment of elementary school students' sun protection behaviors. Pediatr Dermatol. 2010 Mar-Apr;27(2):182-8. doi: 10.1111/j.1525-1470.2009.00940.x. Epub 2009 Jul 20. PMID 19686304
- See also: Information on the Sun protection Project — http://www.safeplay.org